CLINICAL TRIAL: NCT01954706
Title: Pilot Trial of Aerobic and Resistance Exercise Training for the Primary Prevention of Musculoskeletal Side Effects From Aromatase Inhibitors in Postmenopausal Breast Cancer Patients
Brief Title: Exercise to Prevent Aromatase Inhibitor Side Effects in Breast Cancer Patients
Acronym: BCS2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped due to recruitment difficulties
Sponsor: Baltimore VA Medical Center (U.S. Federal Agency)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Susan B. Kesmodel, MD, Assistant Professor of Surgery, Baltimore VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HP-00056384; P30AG028747 (NIH)
Record Dates: First submitted 2013-09-27; First posted 2013-10-07 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Breast Cancer; Sarcopenia
MeSH Terms: conditions — Breast Neoplasms; Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Structured Exercise (Experimental): Structured and supervised aerobic and resistance training 2 times per week
  Interventions: Other: Structured Exercise
- Usual Care (Active Comparator): Subjects will be counseled on American Cancer Society and American College of Sports Medicine physical activity and nutritional guidelines at the initiation of the study. Study participants will be contacted by a physician or nurse on weeks 2, 6, 10, and 14 to provide support and encouragement to patients.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Structured Exercise — Structured and supervised aerobic and resistance training 2 times per week
  Arms: Structured Exercise
Other: Usual Care — Subjects will be counseled on American Cancer Society and American College of Sports Medicine physical activity and nutritional guidelines at the initiation of the study. Study participants will be contacted by a physician or nurse on weeks 2, 6, 10, and 14 to provide support and encouragement to patients.
  Arms: Usual Care

SUMMARY:
Hormone receptor-positive tumors are the most common breast cancers in postmenopausal women, and drug therapies, which block the production or effects of estrogen, are the mainstay of treatment in these patients. Due to their effectiveness in postmenopausal women, aromatase inhibitors (AIs) are the standard of care for long-term estrogen suppression in these patients. Estrogen deficiency, however, results in multiple side effects. Some of the most common side effects in women taking AIs are joint and muscle aches, which promote physical deconditioning. Because of the long term use of AIs in postmenopausal breast cancer patients and the improvements in cancer-related outcomes that are observed with their use, identifying methods to reduce these side effects to maintain adherence to treatment is important. Exercise interventions in breast cancer patients also improve quality of life and reduce fatigue. Understanding the role of exercise in AI side effect prevention will allow us to translate these findings into therapy guidelines.

DETAILED DESCRIPTION:
Breast cancer is the most common malignancy in women in the United States and is the second leading cause of cancer deaths. In 2013, an estimated 230,000 women in the United States will be diagnosed with invasive breast cancer and approximately 40,000 with die.1 Women with breast cancer frequently experience significant functional and metabolic declines during and after treatment due to cancer-related fatigue (CRF), stress and depression.2,3 Cancer-related fatigue is associated with side effects from treatment, pain, functional disability, sleep disturbances, mood disturbances and co-morbid conditions.4 Patients with CRF have declines in physical activity and function, which significantly impacts quality of life (QOL).5 The mechanisms underlying functional declines and fatigue in breast cancer patients are likely multifactorial, but deconditioning, sarcopenia, increases in inflammatory cytokines, insulin resistance, and changes in muscle and fat metabolism seem to play important roles.4,6

Hormone receptor-positive tumors are the most common breast cancers in postmenopausal women, and endocrine therapies, which block the production or effects of estrogen, are the mainstay of treatment in these patients. Due to their superior efficacy in postmenopausal women, aromatase inhibitors (AIs) are the standard of care for long-term estrogen suppression in these patients.7 Estrogen deprivation, however, results in multiple side effects which may worsen fatigue and the functional and metabolic declines associated with cancer treatment.8 Some of the most common side effects in women taking AIs are musculoskeletal symptoms, including arthralgias and myalgias, which promote deconditioning and sarcopenia and their associated side effects.9 Because of the prolonged use of AIs in postmenopausal breast cancer patients and the improvements in cancer-related outcomes that are observed with their use, great efforts are taken to reduce AI induced musculoskeletal symptoms (AIMSS) to maintain adherence to treatment. While multiple strategies are used to manage AIMSS, current therapies mainly focus on interventions in patients who develop symptoms (tertiary prevention) rather than primary prevention.9 Exercise interventions in breast cancer patients also improve QOL, decrease fatigue, and increase physical function and strength.10,11 Understanding the role of exercise in AI side effect prevention will allow us to translate these findings into therapy guidelines.

ELIGIBILITY:
Inclusion Criteria:

* At least mild fatigue in 2 of the 4 areas of the Piper Fatigue Scale (score ≥ 1-3)
* Completion of standard surgery +/- chemotherapy for breast cancer (may undergo radiation therapy during study)
* 25-OH vitamin D > 20 ng/ml
* Histological evidence of stage I-III hormone receptor-positive breast cancer
* Body Mass Index >/=18 and <50 kg/m2
* 40-80 years of age
* Non-smoking (non smoking for at least 12 months: cigarettes, cigars, pipes
* Menopause over one year (absence of menses for 12 months or greater)
* Sedentary (exercise no >60 min 2 times/week)

Exclusion Criteria:

* Taking oral steroids, warfarin, or other medications interfering with fat metabolism that may not be safely discontinued temporarily for specific produces (i.e. for 72 hours prior)
* Symptomatic heart disease, coronary artery disease, congestive heart failure, or uncontrolled hypertension (systolic blood pressure over 180 mm HG)unless medically stabilized
* Participant is, in the opinion of the investigator, unable to adhere to the study protocol due to medical or orthopedic conditions that limit ability to exercise or travel to the Baltimore VA for protocol procedures
* Chronic pulmonary disease (on supplemental O2)
* Abnormal renal function (BUN above 40 mg/dl, Cr above 1.3 mg/dl, CrCl<60mg/dl)
* Unstable lymphedema
* Evidence of cancer metastases or recurrence
* Anemia HCT below 30 mg/dl, platelets below 80,000/cm3
* Type 1 diabetes; insulin treatment for diabetes, poorly controlled diabetes, HgA1c>10%
* Abnormal response to exercise test (ST segment depression greater than 2mm, chest pain, significant arrhythmias, extreme shortness of breath, cyanosis, exercising BP above 240/120 mm HG, or other contraindications to exercise) confirmed with further diagnostic evaluations.
* Abnormal liver function
* Untreated dyslipidemia with National Cholesterol ATPIII 10 year cardiac risk score greater than 10% (www.nhlbi.nih.gov/guidelines/cholesterol/atp3upd04.htm)
* Metal implants or devices (i.e. pacemaker) if undergoing CT scan
* History of seizures or taking anti-seizure or anti convulsion medication
* Allergic to lidocaine
* Mini-mental state examination below 24, dementia, or unstable clinical depression by exam

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-11; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Fatigue | Baseline
  Fatigue (questionnaires) and muscle performance (muscle strength, endurance, and function)
Muscle performance (muscle strength, endurance, and function) Fatigue and Muscle Performance | 16 weeks
  Fatigue (questionnaire) and muscle performance (muscle strength, endurance, and function)
Musculoskeletal symptoms (VASpain, HAQ-DI) | 16 weeks
  Musculoskeletal symptoms (VASpain, HAQ-DI)

SECONDARY OUTCOMES:
Glucose Tolerance and Inflammation | Baseline
Glucose Tolerance and Inflammation | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Susan Kesmodel, MD, Principal Investigator — Baltimore VAMC
Locations (1):
- Baltimore VA Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] Society AC. Cancer Facts & Figures 2013. Atlanta: American Cancer Society 2013.
- [Background] Thomson CA, Thompson PA, Wright-Bea J, Nardi E, Frey GR, Stopeck A. Metabolic syndrome and elevated C-reactive protein in breast cancer survivors on adjuvant hormone therapy. J Womens Health (Larchmt). 2009 Dec;18(12):2041-7. doi: 10.1089/jwh.2009.1365. PMID 20044868
- [Background] Curt GA. Impact of fatigue on quality of life in oncology patients. Semin Hematol. 2000 Oct;37(4 Suppl 6):14-7. doi: 10.1016/s0037-1963(00)90063-5. PMID 11068951
- [Background] Cramp F, Daniel J. Exercise for the management of cancer-related fatigue in adults. Cochrane Database Syst Rev. 2008 Apr 16;(2):CD006145. doi: 10.1002/14651858.CD006145.pub2. PMID 18425939
- [Background] Braithwaite D, Satariano WA, Sternfeld B, Hiatt RA, Ganz PA, Kerlikowske K, Moore DH, Slattery ML, Tammemagi M, Castillo A, Melisko M, Esserman L, Weltzien EK, Caan BJ. Long-term prognostic role of functional limitations among women with breast cancer. J Natl Cancer Inst. 2010 Oct 6;102(19):1468-77. doi: 10.1093/jnci/djq344. Epub 2010 Sep 22. PMID 20861456
- [Background] Berger AM, Gerber LH, Mayer DK. Cancer-related fatigue: implications for breast cancer survivors. Cancer. 2012 Apr 15;118(8 Suppl):2261-9. doi: 10.1002/cncr.27475. PMID 22488700
- [Background] Collado-Hidalgo A, Bower JE, Ganz PA, Cole SW, Irwin MR. Inflammatory biomarkers for persistent fatigue in breast cancer survivors. Clin Cancer Res. 2006 May 1;12(9):2759-66. doi: 10.1158/1078-0432.CCR-05-2398. PMID 16675568
- [Background] Lin NU, Winer EP. Advances in adjuvant endocrine therapy for postmenopausal women. J Clin Oncol. 2008 Feb 10;26(5):798-805. doi: 10.1200/JCO.2007.15.0946. PMID 18258989
- [Background] Dent SF, Gaspo R, Kissner M, Pritchard KI. Aromatase inhibitor therapy: toxicities and management strategies in the treatment of postmenopausal women with hormone-sensitive early breast cancer. Breast Cancer Res Treat. 2011 Apr;126(2):295-310. doi: 10.1007/s10549-011-1351-3. Epub 2011 Jan 20. PMID 21249443
- [Background] Gaillard S, Stearns V. Aromatase inhibitor-associated bone and musculoskeletal effects: new evidence defining etiology and strategies for management. Breast Cancer Res. 2011 Mar 14;13(2):205. doi: 10.1186/bcr2818. PMID 21457526
- [Background] Winters-Stone KM, Dobek J, Bennett JA, Nail LM, Leo MC, Schwartz A. The effect of resistance training on muscle strength and physical function in older, postmenopausal breast cancer survivors: a randomized controlled trial. J Cancer Surviv. 2012 Jun;6(2):189-99. doi: 10.1007/s11764-011-0210-x. Epub 2011 Dec 23. PMID 22193780